CLINICAL TRIAL: NCT05012839
Title: Increased Incidence of Adult Complicated Appendicitis in One Resource-Competent Community During the Coronavirus Disease Pandemic: Time to Improve Health-Seeking Behaviors
Brief Title: Complicated Appendicitis in COVID-19 Era
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202008052RINC
Record Dates: First submitted 2021-08-15; First posted 2021-08-19 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Covid19; Complicated Appendicitis
Keywords: Health-seeking behavior; COVID-19; appendicitis
MeSH Terms: conditions — COVID-19; Health Behavior; Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Complicated appendicitis: The development of complicated appendicitis, diagnosed during appendectomy or by pre-operative image study
  Interventions: Other: impact of COVID-19 on Health-Seeking Behaviors
- Non-complicated appendicitis: No development of complicated appendicitis, diagnosed during appendectomy or by pre-operative image study
  Interventions: Other: impact of COVID-19 on Health-Seeking Behaviors

INTERVENTIONS:
Other: impact of COVID-19 on Health-Seeking Behaviors — The impact of the coronavirus disease 2019 (COVID-19) pandemic on medical services is overwhelming due to limited medical resources. During its initial surge in 2020, Taiwan's government rapidly established diverse public actions, which helped maintain the medical supply without travel restrictions. However, whether the fear of being infected with COVID-19 interfered with health-seeking behavior (HSB) remains unclear. Therefore, this study aimed to elucidate whether acute complicated appendicitis (ACA) rates in adults were affected by the COVID-19 pandemic.

SUMMARY:
Background The impact of the coronavirus disease 2019 (COVID-19) pandemic on medical services is overwhelming due to limited medical resources. During its initial surge in 2020, Taiwan's government rapidly established diverse public actions, which helped maintain the medical supply without travel restrictions. However, whether the fear of being infected with COVID-19 interfered with health-seeking behavior (HSB) remains unclear. Therefore, this study aimed to elucidate whether acute complicated appendicitis (ACA) rates in adults were affected by the COVID-19 pandemic.

Methods A retrospective analysis of acute appendicitis in adults was performed between January 1 and June 30, 2020 (COVID-19 period). The control period was collected from the first two quarters for the preceding 3 years. Outcome measures were ACA and length of hospital stays.

ELIGIBILITY:
Inclusion Criteria:

* Acute appendicitis

Exclusion Criteria:

* No

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A retrospective analysis of acute appendicitis in adults was performed between January 1 and June 30, 2020 (COVID-19 period). The control period was collected from the first two quarters for the preceding 3 years. Outcome measures were ACA and length of hospital stays.
Sampling Method: Non-Probability Sample
Enrollment: 465 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-08-14 (Actual)

PRIMARY OUTCOMES:
Incidence of complicated appendicitis | baseline, pre-surgery
  The primary outcome measure was the occurrence of ACA defined as abscess observed in computed tomography, presence of appendiceal perforation determined by surgical documentation, or a description of gangrenous appendicitis assessed by pathological reports.

SECONDARY OUTCOMES:
Length of hospital stays | up to 4 weeks
  the duration of hospital stays after surgery

IPD SHARING:
Plan to Share IPD: No